CLINICAL TRIAL: NCT02611648
Title: Prospective Randomized Double-blinded Trial Comparing Three Duodenoscope High- Level Disinfection and Sterilization Procedures
Brief Title: Duodenoscope Disinfect Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Mandeep Sawhney, Mandeep Sawhney, MD, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2015P000263
Record Dates: First submitted 2015-11-12; First posted 2015-11-23 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Endoscopic Retrograde Cholangiopancreatogram (ERCP)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- standard HLD (No Intervention): Standard high-level disinfectant (metricide ortho-phthalaldehyde) currently performed at BIDMC (standard HLD)
- double HLD (Experimental): Double the exposure time of the standard high level disinfectant (metricide ortho-phthalaldehyde)
  Interventions: Other: Double HLD
- HLD/ETO (Experimental): Standard high level disinfectant (metricide ortho-phthalaldehyde) followed by ethylene oxide
  Interventions: Other: HLD/ETO

INTERVENTIONS:
Other: Double HLD — Standard high level disinfectant (metricide ortho-phthalaldehyde) with an additional exposure time to disinfect
  Arms: double HLD
Other: HLD/ETO — Standard high level disinfectant (metricide ortho-phthalaldehyde) followed by ethylene oxide
  Arms: HLD/ETO

SUMMARY:
This study is investigating the most effective way to sterilize duodenoscopes ("scopes") used at Beth Israel Deaconess Medical Center (BIDMC). Right now, BIDMC uses the standard method of high level disinfection to sterilize scopes. Because infections have been passed by scopes at other institutions in the U.S., the investigators are exploring whether or not adding two different sterilization processes will reduce this risk of contamination.

Bacteria may be passed from a patient's intestines to the scope. Or, if the scope is contaminated, bacteria may be passed from the scope to the patient. In order to understand how bacteria are passed, the investigators will be taking samples of the patient's intestinal bacteria to compare to the bacteria, if any, found on the scope.

DETAILED DESCRIPTION:
Study Design

This study is designed to evaluate the effect of supplementing standard high-level disinfection with additional high level-disinfection or sterilization procedures on the frequency of duodenoscopes contamination. Duodenoscopes will be randomly assigned to one of three arms:

* Standard high-level disinfection currently performed at BIDMC (standard HLD)
* Standard high-level disinfection with an additional exposure time to disinfectant (double HLD)
* Standard high-level disinfection followed by ethylene oxide (HLD/ETO)

The study will be conducted with the following elements:

1. All duodenoscopes will be randomly assigned to a study arm before the duodenoscope is used for an Endoscopic Retrograde Cholangiopancreatogram (ERCP) procedure included in the study, including duodenoscopes introduced during the study.
2. All duodenoscopes used for ERCP will have the following cultures obtained in a sterile fashion
3. Patient study consent for obtaining patient rectal surveillance and clinical cultures will be obtained at the time of ERCP procedure consent among all patients undergoing ERCP. Patients will be blinded to duodenoscope disinfection/sterilization assignment.
4. The ERCP procedure will be performed according to standard clinical practice. Among patients consenting to specimen collection, a duodenal aspirate will be obtained during the procedure.
5. Among consenting patients, a rectal surveillance swab will be collected post-procedurally by ERCP staff.
6. After ERCP completion, current BIDMC-employed trained technicians will perform the assigned disinfection/sterilization procedure.

ELIGIBILITY:
Inclusion Criteria:

1. A duodenoscope used for any intended ERCP procedure will be included in the study
2. All adult patients (age ≥18 years) scheduled to undergo ERCP will be offered participation in patient specimen collection component of the study

Exclusion Criteria:

1. Patients in whom ERCP or endoscopy with a duodenoscope is medically contra-indicated will not be included in the patient specimen collection portion of the study
2. Patients with surgically altered anatomy in whom ERCP is performed using an enteroscope (and not a duodenoscope) will not be included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 541 (Actual)
Dates: Start 2015-11; Primary Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Frequency of contaminated duodenoscopes after using three different types of disinfection processes | 6 months
  Compare the frequency of duodenoscope contamination after reprocessing using 3 different methods: standard high-level disinfection procedure with ortho-phthalaldehyde (standard HLD), double cycle of standard high-level disinfection (double HLD), and standard high-level disinfection followed by ethylene oxide (ETO) gas sterilization (HLD/ETO)

REFERENCES:
- [Derived] Snyder GM, Wright SB, Smithey A, Mizrahi M, Sheppard M, Hirsch EB, Chuttani R, Heroux R, Yassa DS, Olafsdottir LB, Davis RB, Anastasiou J, Bapat V, Bidari K, Pleskow DK, Leffler D, Lane B, Chen A, Gold HS, Bartley A, King AD, Sawhney MS. Randomized Comparison of 3 High-Level Disinfection and Sterilization Procedures for Duodenoscopes. Gastroenterology. 2017 Oct;153(4):1018-1025. doi: 10.1053/j.gastro.2017.06.052. Epub 2017 Jul 13. PMID 28711629